CLINICAL TRIAL: NCT05047445
Title: A First Time in Human Phase 1 Open-Label Study of the Safety, Tolerability, and Immunogenicity of COVIDITY Vaccine Administered by Needle-free Intradermal Injection or Needle-free Intramuscular Injection in Healthy Adults (COVIDITY-001)
Brief Title: A First Time in Human Phase 1 Open-Label Study of the COVIDITY Vaccine Administered by Needle-free Injection
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Scancell Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: COVIDITY-001
Record Dates: First submitted 2021-08-27; First posted 2021-09-17 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Open label, uncontrolled study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COVIDITY administered via needle-free intradermal injection (PharmaJet Tropis) (Experimental)
  Interventions: Biological: COVIDITY (SCOV1 and SCOV2) administered via needle-free intradermal injection; Biological: COVIDITY (SCOV2 only) administered via needle-free intradermal injection to vaccine naive and/or previously vaccinated participants; Biological: COVIDITY (SCOV2 only) administered via needle-free intradermal injection to previously infected participants
- COVIDITY administered via needle-free intramuscular injection (PharmaJet Stratis) (Experimental)
  Interventions: Biological: COVIDITY (SCOV1 and SCOV2) administered via needle-free intramuscular injection; Biological: COVIDITY (SCOV2 only) administered via needle-free intramuscular injection to vaccine naive and/or previously vaccinated participants; Biological: COVIDITY (SCOV2 only) administered via needle-free intramuscular injection to previously infected participants

INTERVENTIONS:
Biological: COVIDITY (SCOV1 and SCOV2) administered via needle-free intradermal injection — Two 0.2 mg doses of the plasmid DNA vaccine SCOV1 (administered on Day 1 and Day 29), followed by two 0.2 mg doses of the plasmid DNA vaccine SCOV2 (not before Days 113 and 141 [doses 4 weeks apart]).
  Arms: COVIDITY administered via needle-free intradermal injection (PharmaJet Tropis)
Biological: COVIDITY (SCOV1 and SCOV2) administered via needle-free intramuscular injection — Two 1.0 mg doses of the plasmid DNA vaccine SCOV1 (administered on Day 1 and Day 29), followed by two 1.0 mg doses of the plasmid DNA vaccine SCOV2 (not before Days 113 and 141 [doses 4 weeks apart]).
  Arms: COVIDITY administered via needle-free intramuscular injection (PharmaJet Stratis)
Biological: COVIDITY (SCOV2 only) administered via needle-free intradermal injection to vaccine naive and/or previously vaccinated participants — Two 0.8 mg doses of the plasmid DNA vaccine SCOV2 administered on Day 1 and Day 29
  Arms: COVIDITY administered via needle-free intradermal injection (PharmaJet Tropis)
Biological: COVIDITY (SCOV2 only) administered via needle-free intramuscular injection to vaccine naive and/or previously vaccinated participants — Two 4.0 mg doses of the plasmid DNA vaccine SCOV2 administered on Day 1 and Day 29
  Arms: COVIDITY administered via needle-free intramuscular injection (PharmaJet Stratis)
Biological: COVIDITY (SCOV2 only) administered via needle-free intradermal injection to previously infected participants — A single 0.8 mg dose of the plasmid DNA vaccine SCOV2 administered on Day 1
  Arms: COVIDITY administered via needle-free intradermal injection (PharmaJet Tropis)
Biological: COVIDITY (SCOV2 only) administered via needle-free intramuscular injection to previously infected participants — A single 4.0 mg dose of the plasmid DNA vaccine SCOV2 administered on Day 1
  Arms: COVIDITY administered via needle-free intramuscular injection (PharmaJet Stratis)

SUMMARY:
The main objectives of this study are to assess the safety, tolerability and immunogenicity of the candidate SARS-CoV-2 vaccine, COVIDITY, when administered using a needle-free ID or IM injection device.

DETAILED DESCRIPTION:
This is a first time in human (FTiH) study designed to explore the safety, tolerability, and immunogenicity of COVIDITY in healthy adults when administered by needle-free injection.

COVIDITY consists of two DNA plasmid vaccines (SCOV1 and SCOV2). SCOV1 is expected to be active against the original SARS-CoV-2 strain and the B.1.1.7 (Alpha) variant, and to a slightly lesser extent against the B.1.351 (Beta) and P.1 (Gamma) variants. SCOV2 is expected to boost the effects of SCOV1 while providing further enhanced protection against the B.1.351 (Beta) and P.1 (Gamma) variants. Antibodies induced by SCOV1 and SCOV2 also show strong binding to the B.1.617.2 (Delta) and B.1.1.529 (Omicron) variants in nonclinical models.

When the study commenced in 2021 there were significant numbers of unvaccinated individuals who also had no known exposure to SARS-CoV-2; however as the epidemiology rapidly changed with most people having either been vaccinated, or infected with SARS-CoV-2, or both, the use of SCOV2 only in these populations made rational sense, particularly as it has more mutations in common with the Omicron variant. A protocol amendment submitted in February 2022, permitted the enrolment of participants irrespective of their previous COVID-19 vaccination and/or SARS-CoV-2 infection status, amended the treatment regimen to SCOV2 only, and aligned the administered dose with the doses employed for other DNA vaccines. Immunogenicity analyses will be performed separately for the vaccine-naïve, previously vaccinated and previously infected immunogenicity analysis populations.

Eligible participants will be randomised 1:1 to be vaccinated by either IM or ID needle-free injection in blocks determined by their previous COVID-19 vaccination and SARS-CoV-2 infection status, as follows:

Participants enrolled under the initial protocol (Amendment 1): Two doses of SCOV1 (administered on Day 1 and Day 29), followed by two doses of SCOV2 (not before Days 113 and 141 [doses 4 weeks apart]). A final end of study assessment will then be performed 6 weeks after last dose of study vaccine (Day 183).

Participants enrolled under protocol Amendment 2: Vaccine Naive and Previously Vaccinated participants: Two doses of SCOV2 (administered on Day 1 and Day 29) with a final end of study assessment performed 6 weeks after last dose of study vaccine (Day 71); Previously Infected participants: A single dose of SCOV2 (administered on Day 1) with a final end of study assessment performed 6 weeks after last dose of study vaccine (Day 43)

Each dose of SCOV1 and/or SCOV2 will be administered via needle-free injection, either intradermally (study Arm 1; PharmaJet Tropis® device) or intramuscularly (study Arm 2; PharmaJet Stratis® device). Eligible injection sites include the outer aspect of the upper left or right arm (medial deltoid muscle) or the left or right outer thigh (lateralis muscle).

This study is expected to enrol up to 80 participants at a single centre in South Africa. Enrolment will attempt to continue until at least 10 evaluable participants receive all protocol-required SCOV2 vaccinations for each immunogenicity analysis population. However, should the epidemiology be such that certain populations cannot be enrolled, the Safety Review Committee may determine that enrolment for that population be considered complete.

ELIGIBILITY:
Participants must meet ALL of the following Inclusion Criteria to be eligible for study entry:

* Participant is able and willing to provide written informed consent prior to any study procedure.
* Participant is 18 to 59 years of age.
* Participant is male or non-pregnant female.
* Participant has had no known exposure to SARS-CoV-2 virus in the last 14 days and has a negative RT-PCR SARS-CoV-2 laboratory test within 48 hours prior to the first study vaccination administration.
* Participant is determined by the Investigator to be healthy on the basis of medical history, physical examination, vital signs, and routine laboratory tests.
* Participant agrees to comply with study procedures, including the collection of venous blood, and to be available for all study visits.
* Women of child-bearing potential must have a negative urine pregnancy test during screening and a negative serum pregnancy test on Day -1, prior to the first dose of study vaccine, and be neither breastfeeding nor intending to become pregnant during study participation. Women of child-bearing potential must agree to use highly effective contraceptive methods at least 28 days prior to study entry, for the duration of study participation, and for 120 days after the last dose of study vaccine
* Men who are potentially fertile must agree to use barrier protection for the duration of their participation in the study and until 120 days after administration of the last dose of study vaccine when they engage in sexual relations with women who are of child-bearing potential, pregnant, or lactating; they also agree to request their female partners to use an effective method of contraception if they are of child-bearing potential
* Participant has an oral temperature of less than 37.5 oC at screening and prior to dosing.
* Participant has a screening electrocardiogram (ECG) with none of the following clinically significant findings:

  * PR-interval >210 msec
  * QRS-duration >120 msec
  * QT-interval >500 msec
  * Corrected QT-interval by Fridericia (QTcF)-interval >450 msec (males), >470 msec (females)
  * Pathologic Q wave
  * Significant ST-T wave changes
  * Second or third-degree atrioventricular heart block.
* Participant agrees to refrain from donating blood or plasma, outside of the study, for the duration of study participation, and for 28 days after the last dose of study vaccine.
* Participant agrees not to consume any alcohol within 48 hours prior to each study vaccine administration and has a negative alcohol breath test prior to the first administration of the study vaccine.

Participant's meeting ANY of the following Exclusion Criteria are not eligible for study entry:

* Participant has a history of proven infection with SARS-CoV-2 during the 28 days prior to the first planned administration of COVIDITY.
* Participant has received a COVID-19 or other vaccination or booster during the 28 days prior to the first planned administration of COVIDITY.
* Participant has a history of chronic respiratory disease, hypertension, significant cardiovascular disease, autoimmune disease (including hypothyroidism without defined non-autoimmune cause), immunodeficiency, clotting disorder, history of thrombosis, or malignancy (except for adequately treated malignancies with an expected 5-year survival rate of >90%, e.g., carcinoma in-situ of the breast or cervix, squamous or basal cell carcinoma of the skin).
* Participant has any medical disease or condition, or psychiatric condition, which in the opinion of the Investigator would preclude study participation (would place the participant at an unacceptable risk of injury, render the participant unable to meet the requirements of the protocol, or may interfere with the evaluation of responses).
* Participant has a positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus types 1 or 2 antibodies at screening.
* Alcohol consumption of >21 units per week (males) or >14 units per week (females) (1 unit of alcohol equals 1/2 pint [285 mL] of beer or lager, 1 glass [125 mL] of wine, or 1/6 gill [25 mL] of spirits).
* History of strenuous exercise (e.g., heavy lifting, weight, or fitness training) within 96 hours (4 days) prior to administration of the first study vaccination.
* Participant has participated in another investigational study involving an investigational product within 30 days, or 5 half-lives, whichever is longer, before the first study vaccine administration in the current study.
* Participant is currently enrolled in or plans to participate in another clinical trial with an investigational product that will be received during the study reporting period.
* Participant has a history of any vaccine or drug hypersensitivity reactions (including skin reactions or anaphylaxis), or other known clinically significant allergies.
* Participant has a history of chronic use (>14 continuous days in the 6 months preceding screening) of any medications that may be associated with impaired immune responsiveness including, but not limited to: systemic corticosteroids exceeding 10 mg/day of prednisone equivalent, allergy injections, immunoglobulin, interferon, immunomodulators, cytotoxic drugs, or other immuno-suppressive drugs. The use of low dose topical, ophthalmic, inhaled, and intranasal steroid preparations is permitted (not more than the equivalent of 10 mg prednisone a day).
* Use of any prescription medications within 14 days or 5 half-lives (whichever is longer) of first study vaccine administration (Day 1), use of over-the-counter medications or herbal supplements within 7 days. The use of occasional paracetamol (up to 4 g per day) and hormone replacement therapy, oral, implantable, transdermal injectable or intrauterine contraceptives is permitted. Nutritional supplements may be permitted but must be discussed with the Sponsor's medical monitor prior to participant enrolment.
* Participant has received immunoglobulins and/or any blood or blood products within 90 days before the first study vaccine administration (Day 1) or at any time during the study.
* Participant has a history of alcohol abuse or other recreational drug (excluding cannabis) use within 6 months before the first study vaccine administration.
* Participant has a positive result for urine drugs of abuse at screening or prior to the first study vaccine administration (Day 1) with the exception of cannabis for which a positive result is acceptable if the participant confirms recreational use, and this information is considered to be reliable in the opinion of the Investigator.
* Participant has received an experimental SARS-CoV-2 vaccine other than SCOV1.
* Participant is pregnant, lactating, or is planning or wanting to conceive/father children during the study.
* Participant has any clinically significant abnormal findings on screening biochemistry, haematology or coagulation blood tests, or urinalysis; participants with Gilbert's syndrome will be permitted to enter the study.
* Any other reason that, in the opinion of the Investigator, may render the participant unable to participate in the study, may limit their ability to provide participant reported outcomes, or may interfere with protocol adherence.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of COVIDITY as assessed by the recording of adverse events (AEs) | From enrolment through end of study; approximately 6 to 26 weeks
  National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events; CTCAE v5.0.
Safety and tolerability of COVIDITY as assessed by the recording of vital signs | From enrolment through end of study; approximately 6 to 26 weeks
  Oral temperature (°C)
Safety and tolerability of COVIDITY as assessed by the recording of vital signs | From enrolment through end of study; approximately 6 to 26 weeks
  Pulse (beats per minute)
Safety and tolerability of COVIDITY as assessed by the recording of vital signs | From enrolment through end of study; approximately 6 to 26 weeks
  Respiratory rate (breaths per minute)
Safety and tolerability of COVIDITY as assessed by the recording of vital signs | From enrolment through end of study; approximately 6 to 26 weeks
  Systolic and diastolic blood pressure (mm Hg)
Safety and tolerability of COVIDITY as assessed by a physical examination of the participant | From enrolment through end of study; approximately 6 to 26 weeks
  Physical examination findings (binary classification: normal or abnormal)
Safety and tolerability of COVIDITY as assessed by serum chemistry | From enrolment through end of study; approximately 6 to 26 weeks
  Albumin (g/L)
Safety and tolerability of COVIDITY as assessed by serum chemistry | From enrolment through end of study; approximately 6 to 26 weeks
  Alanine aminotransferase (IU/L)
Safety and tolerability of COVIDITY as assessed by serum chemistry | From enrolment through end of study; approximately 6 to 26 weeks
  Alkaline phosphatase (IU/L)
Safety and tolerability of COVIDITY as assessed by serum chemistry | From enrolment through end of study; approximately 6 to 26 weeks
  Aspartate aminotransferase (IU/L)
Safety and tolerability of COVIDITY as assessed by serum chemistry | From enrolment through end of study; approximately 6 to 26 weeks
  Bicarbonate (mmol/L)
Safety and tolerability of COVIDITY as assessed by serum chemistry | From enrolment through end of study; approximately 6 to 26 weeks
  Corrected Calcium (mmol/L).
Safety and tolerability of COVIDITY as assessed by serum chemistry | From enrolment through end of study; approximately 6 to 26 weeks
  Chloride (mmol/L)
Safety and tolerability of COVIDITY as assessed by serum chemistry | From enrolment through end of study; approximately 6 to 26 weeks
  Creatinine (μmol/L)
Safety and tolerability of COVIDITY as assessed by serum chemistry | From enrolment through end of study; approximately 6 to 26 weeks
  Creatine kinase (IU/L)
Safety and tolerability of COVIDITY as assessed by serum chemistry | From enrolment through end of study; approximately 6 to 26 weeks
  Total bilirubin (and direct if clinically indicated; μmol/L)
Safety and tolerability of COVIDITY as assessed by serum chemistry | From enrolment through end of study; approximately 6 to 26 weeks
  Gamma glutamyl transferase (IU/L)
Safety and tolerability of COVIDITY as assessed by serum chemistry | From enrolment through end of study; approximately 6 to 26 weeks
  Lactate dehydrogenase (IU/L)
Safety and tolerability of COVIDITY as assessed by serum chemistry | From enrolment through end of study; approximately 6 to 26 weeks
  Random glucose (mmol/L)
Safety and tolerability of COVIDITY as assessed by serum chemistry | From enrolment through end of study; approximately 6 to 26 weeks
  Phosphorus (measured as phosphate; mmol/L)
Safety and tolerability of COVIDITY as assessed by serum chemistry | From enrolment through end of study; approximately 6 to 26 weeks
  Potassium (mmol/L)
Safety and tolerability of COVIDITY as assessed by serum chemistry | From enrolment through end of study; approximately 6 to 26 weeks
  Sodium (mmol/L)
Safety and tolerability of COVIDITY as assessed by serum chemistry | From enrolment through end of study; approximately 6 to 26 weeks
  Uric acid (urate; mmol/L)
Safety and tolerability of COVIDITY as assessed by serum chemistry | From enrolment through end of study; approximately 6 to 26 weeks
  Total protein (g/L)
Safety and tolerability of COVIDITY as assessed by haematology | From enrolment through end of study; approximately 6 to 26 weeks
  Haemoglobin (g/dL)
Safety and tolerability of COVIDITY as assessed by haematology | From enrolment through end of study; approximately 6 to 26 weeks
  Haematocrit (L/L)
Safety and tolerability of COVIDITY as assessed by haematology | From enrolment through end of study; approximately 6 to 26 weeks
  Mean corpuscular volume (fL)
Safety and tolerability of COVIDITY as assessed by haematology | From enrolment through end of study; approximately 6 to 26 weeks
  Mean corpuscular haemoglobin concentration (g/dL)
Safety and tolerability of COVIDITY as assessed by haematology | From enrolment through end of study; approximately 6 to 26 weeks
  Platelet count (cells x 10^9/L)
Safety and tolerability of COVIDITY as assessed by haematology | From enrolment through end of study; approximately 6 to 26 weeks
  Red blood cell count (cells x 10^12/L)
Safety and tolerability of COVIDITY as assessed by haematology | From enrolment through end of study; approximately 6 to 26 weeks
  White blood cell count (cells x 10^9/L)
Safety and tolerability of COVIDITY as assessed by haematology | From enrolment through end of study; approximately 6 to 26 weeks
  White blood cell differential (cells x 10^9/L)
Safety and tolerability of COVIDITY as assessed by coagulation parameters and biomarkers | From enrolment through end of study; approximately 6 to 26 weeks
  International normalised ratio (no units)
Safety and tolerability of COVIDITY as assessed by coagulation parameters and biomarkers | From enrolment through end of study; approximately 6 to 26 weeks
  Activated partial prothrombin time (sec)
Safety and tolerability of COVIDITY as assessed by coagulation parameters and biomarkers | From enrolment through end of study; approximately 6 to 26 weeks
  Fibrinogen (g/L)
Safety and tolerability of COVIDITY as assessed by coagulation parameters and biomarkers | From enrolment through end of study; approximately 6 to 26 weeks
  D-dimer (ng/mL)
Safety and tolerability of COVIDITY as assessed by urinalysis | From enrolment through end of study; approximately 6 to 26 weeks
  Glucose (negative, 100/250/500/1000/2000+ mg/dL)
Safety and tolerability of COVIDITY as assessed by urinalysis | From enrolment through end of study; approximately 6 to 26 weeks
  Ketones (negative, trace/small/moderate/large, 5/15/40/80/160 mg/dL)
Safety and tolerability of COVIDITY as assessed by urinalysis | From enrolment through end of study; approximately 6 to 26 weeks
  Blood (negative, trace, non-haemolysed trace/moderate, haemolysed trace/+/++/+++)
Safety and tolerability of COVIDITY as assessed by urinalysis | From enrolment through end of study; approximately 6 to 26 weeks
  Leucocytes (negative, trace/+/++/+++)
Safety and tolerability of COVIDITY as assessed by urinalysis | From enrolment through end of study; approximately 6 to 26 weeks
  Bilirubin (negative, +/++/+++)
Safety and tolerability of COVIDITY as assessed by urinalysis | From enrolment through end of study; approximately 6 to 26 weeks
  pH (5.0/5.5/6.0/6.5/7.0/7.5/8.0/8.5 pH units)
Safety and tolerability of COVIDITY as assessed by urinalysis | From enrolment through end of study; approximately 6 to 26 weeks
  Specific gravity (1.000/1.004/1.005/1.010/1.015/1.020/1.025/1.030 [no units])
Safety and tolerability of COVIDITY as assessed by urinalysis | From enrolment through end of study; approximately 6 to 26 weeks
  Protein (negative, trace/+/++/+++/++++)
Safety and tolerability of COVIDITY as assessed by urinalysis | From enrolment through end of study; approximately 6 to 26 weeks
  Microscopy (if clinically indicated only) examination for bacteria, red blood cells, white blood cells, casts, and crystals (binary classification: absent or present)
Safety and tolerability of COVIDITY as assessed by 12-lead electrocardiogram (ECG) | From enrolment through end of study; approximately 6 to 26 weeks
  Heart rate, PR-interval, QRS-duration, QT-interval, corrected QT-interval by Fridericia (QTcF), general morphology, and the interpretation of the ECG by the Investigator
Safety and tolerability of COVIDITY as assessed by local and systemic reactogenicity events | From enrolment through end of study; approximately 6 to 26 weeks
  Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (US FDA 2007).
  Local reactogenicity events will be measured for the injection site using a 4-point scale where 1 = 'mild' and 4 = 'potentially life-threatening'.
  Systemic reactogenicity events of interest include fever, chills, headache, myalgia, arthralgia, fatigue, nausea, vomiting, diarrhoea, rhinorrhoea, wheezing, general feeling of being unwell, and loss of appetite.
Safety and tolerability of COVIDITY as assessed by the onset of any new chronic medical conditions | From enrolment through end of study; approximately 6 to 26 weeks

SECONDARY OUTCOMES:
The immunogenicity of COVIDITY as assessed by antibody response | From enrolment through end of study; approximately 6 to 26 weeks
  Quantitative COVIDITY-specific antibody responses measured by enzyme-linked immunosorbent assay (ELISA) or using the Meso Scale Discovery (MSD) platform
The immunogenicity of COVIDITY as assessed by seroconversion and/or increase in antibody titre | From enrolment through end of study; approximately 6 to 26 weeks
  The proportion of participants who seroconvert and/or have a 4-fold increase in N ± S protein antibody titre from baseline
The immunogenicity of COVIDITY as assessed by T cell response | From enrolment through end of study; approximately 6 to 26 weeks
  Quantitative COVIDITY-specific T cell responses measured by ELISpot assay

OTHER OUTCOMES:
Exploratory: The proportion of participants who remain COVID-19 free throughout the study | From enrolment through end of study; approximately 6 to 26 weeks
  The proportion of participants that remain negative for the SARS-CoV-2 reverse transcriptase polymerase chain reaction (RT-PCR) test throughout the duration of the study
Exploratory: The induction of a functional humoral immune response by COVIDITY | From enrolment through end of study; approximately 6 to 26 weeks
  Pseudovirus neutralisation assay, live virus neutralisation assay or angiotensin converting enzyme 2 (ACE2) neutralisation assay Analysis of immune responses in participants who are SARS-CoV-2 positive.
Exploratory: The induction of a functional humoral immune response by COVIDITY | From enrolment through end of study; approximately 6 to 26 weeks
  c) Analysis of immune responses using intracellular staining, immune cell phenotyping by flow cytometry, cytotoxicity assays, proliferation assay, cytokine analysis, tetramer staining, and T cell receptor repertoire analysis

CONTACTS AND LOCATIONS:
Overall Officials: Rodney Dawson, MD, Principal Investigator — University of Cape Town Lung Institute
Locations (1):
- University of Cape Town Lung Institute, Centre for TB Research Innovation, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual patient data available.